CLINICAL TRIAL: NCT03744481
Title: Becoming Children With Perinatal Anoxo-Ischemic Encephalopathy Without Indication of Therapeutic Hypothermia
Acronym: SARNATUN
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0627
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Anoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionaire — Evaluation of psychomotor development in children with mild EAI without indication of therapeutic hypothermia.
  Precise analysis of the type (motor, sensory, language, epilepsy) and the severity of sequelae by sending a questionnaire to parents.
  Investigation of early, clinical and paraclinical prognostic factors of good or bad neurodevelopmental outcome.
  Evaluation of the height-weight growth and the cranial perimeter

SUMMARY:
There are 3 levels of severity of anoxo-ischemic encephalopathy (EAI): mild, moderate and severe. Therapeutic hypothermia is beneficial in children with moderate EAI. It is ineffective in severe EAI and may be deleterious if there is no EAI. He continues to question his interest in light EAIs.

There are few studies on the becoming of children with a mild anoxic-ischemic encephalopathy and not set hypothermia.

The main hypothesis of the study is that term newborns with anoxo-ischemic encephalopathy who did not require therapeutic hypothermia have normal psychomotor development at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Full-term children, gestational age> 36 weeks of amenorrhea
* Between the 1st of January 2012 and the 31st of December 2016
* Hospitalized in the neonatal resuscitation department of Croix Rousse in Lyon
* Perinatal asphyxia with clinical signs of encephalopathy
* Indication of therapeutic hypothermia not retained because EAI mild
* Where parents were informed and did not object to participation in the study

Exclusion Criteria:

* Dysmorphic syndrome
* Stroke
* Children transferred for other criteria (respiratory distress, heart failure ...)

Ages: 2 Years to 7 Years | Sex: All
Age Groups: Child
Study Population: Full term children with perinatal asphyxia and with clinical signs of mild EAI without indication of therapeutic hypothermia
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-05-19 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Existence of abnormalities | maximum 1 years
  Abnormalities researched are : abnormal motor, sensory (auditory or visual), delayed psychomotor acquisition compared to the expected (norms), or epilepsy at 2 years.
  These anomalies will be collected by sending a questionnaire to the parents.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation néonatale - Hôpital de la Croix Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No